CLINICAL TRIAL: NCT00175084
Title: Effect of Dietary Amino Acid Profile on Lipoprotein Metabolism, Vascular Reactivity and Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HL58008-1188
Record Dates: First submitted 2005-09-08; First posted 2005-09-15 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Hyperlipidemias; Metabolic Syndrome X; Cardiovascular Diseases
MeSH Terms: conditions — Hyperlipidemias; Metabolic Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Comparison of dietary protein amino acid profile — Healthy adults over 50 years of age (men and postmenopausal women) will be assigned to one of two diets differing in lysine to arginine ration (0.7 vs. 1.4) for a 5 week period and then switched to the alternate diet, with a 2 to 4-week washout period, in a randomized crossover design. Blood samples will be collected three times in the fasted state and once 4-hours after the evening meal during the last week of each dietary period of measurement of concentration of plasma lipids, lipoproteins, apolipoproteins, arginine, C-reactive protein, nitrites/nitrates, homocysteine, lecithin-cholesterol acetyltransferase (LCAT), cholesteryl ester transfer protein (CETP), and LDL-receptor messenger ribonucleic acid (mRNA) expression.A 24-hour urine sample will be collected at the end of each phase to measure F2-isoprostanes as an indicator of whole body oxidation.

SUMMARY:
The aim of this study is to explore the significance of the Lys:Arg ratio on responses of lipids and lipoprotein concentrations to dietary proteins and to evaluate the effects of dietary Lys:Arg on cardiovascular disease risk factors and endothelial function.

DETAILED DESCRIPTION:
Findings from early studies in a variety of experimental models of atherosclerosis on the effect of dietary protein suggested that proteins from vegetable sources are less cholesterolemic and atherogenic than proteins from animal sources. Throughout the later part of the 20th century there has been sporadic interest in the effect of protein type and amino acid profiles on blood lipid concentrations and atherosclerosis. A major focus for this evaluation has been to compare proteins based on their amino acid profile, often expressed as lysine (Lys) to arginine (Arg) ratio (Lys:Arg). While animal studies have provided important information regarding the significance of the Lys:Arg in determining the cholesterolemic response to a dietary protein, interpretation of these data must be done with caution since most of the studies have been conducted in animal models that have a different lipoprotein distribution and metabolism than humans. Moreover, the mechanistic insights of this response are yet to be determined. While the favorable effects of Arg on endothelial function appear to be consistent when Arg is administered using a supplement, the effects of dietary Arg naturally present in protein rich foods has yet to be determined. The aim of this proposal is to explore the significance of the Lys:Arg ratio on responses of lipids and lipoprotein concentrations to dietary proteins and to evaluate the effects of dietary Lys:Arg on cardiovascular disease risk factors and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-85 years
* LDL-C concentrations >120 mg/dL

Exclusion Criteria:

* Use of medications known to affect lipid metabolism
* Established cardiovascular disease
* Renal disease
* Liver disease
* Thyroid disease unless controlled with medication for at least 6 months
* Type I and II diabetes
* Irritable bowel syndrome
* Chronic use of prescription anti-inflammatory medications
* Smoking
* Alcohol intake >7 alcoholic drinks per week
* Unwillingness to maintain body weight during participation in the study
* triglyceride (TG) > 400 mg/dL
* Unwillingness to adhere to diet and study protocol
* Weight gain or loss of more than 15 lb within 6 months prior to enrollment

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-10; Primary Completion 2007-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Serum lipid and lipoprotein concentrations, endothelial function, blood pressure, indicators of nitrous oxide end products, homocysteine, inflammation and oxidation markers. | 5 week

CONTACTS AND LOCATIONS:
Overall Officials: Alice H Lichtenstein, D.Sc., Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- See also: Click here for more information about this study: — http://hnrc.tufts.edu